CLINICAL TRIAL: NCT03724058
Title: Fixation and Stability of the Trident® II Clusterhole HA Shells Compared to the Trident® Hemi HA Shells With X3. A Single Center RSA Study
Brief Title: Fixation and Stability of the Trident® II Clusterhole HA Shells
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-I-104
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Hip Replacement Arthroplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Trident® II Clusterhole HA Acetabular Shell (Experimental): Hip arthroplasty using Trident II Clusterhole HA Acetabular Shells
  Interventions: Device: Trident® II Clusterhole HA Acetabular Shell
- Trident® Hemispherical Acetabular Shell (Active Comparator): Hip arthroplasty using Trident Hemispherical Acetabular Shell
  Interventions: Device: Trident® Hemispherical Acetabular Shell

INTERVENTIONS:
Device: Trident® II Clusterhole HA Acetabular Shell — Hip arthroplasty
  Other Names: Stryker Orthopaedics
  Arms: Trident® II Clusterhole HA Acetabular Shell
Device: Trident® Hemispherical Acetabular Shell — Hip arthroplasty
  Other Names: Stryker Orthopaedics
  Arms: Trident® Hemispherical Acetabular Shell

SUMMARY:
The purpose of the Trident® II project is to introduce a cup system that modernizes and streamlines Stryker's acetabular shell portfolio. The Trident® II Clusterhole HA Shell combines the history of Stryker's Trident® shells with plasma spray CpTi with HA coating. Plasma spray coating and HA is considered to be the gold standard in orthopaedics today. This coating will help the cup to achieve early stability and long term fixation.

One of the causes for implant failure is loosening and osteolysis. Osteolysis can be triggered when metal or polyethylene wear particles from the implant or bearing surfaces migrate between implant and surrounding host bone tissue. With the development of sequential irradiated and annealed highly crosslinked polyethylene (X3) wear rates (mean proximal, 2-dimensional and 3-dimensional) have been substantially reduced to 0.001 mm/y, calculated between 1 year and 5 years.

The Trident® II Clusterhole HA shells have a plasma sprayed CpTi coating compared to the arc-deposition CpTi coating on legacy Trident® shells, both designed to allow bone ongrowth. With this study the investigators want to prove equivalent implant fixation of both type of cups.

The primary objective is the assessment of prosthetic fixation and migration results after two years of the Trident® II Clusterhole HA shell compared to the legacy Trident® Hemi HA shell by means of RSA. It is hypothesized that they will perform equally.

The secondary outcome measure will be long-term (10-year) survival based on the two-year migration patterns combined with clinical factors and radiographic aspects. In order to identify other clinical parameters besides the fixation of the prosthesis components, clinical scores and radiographic aspects will be correlated with the RSA outcome. The 10-year results will be used to verify the predicted long-term survival results.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to understand the meaning of the study and is willing to sign the EC approved, study specific Informed Patient Consent Form.
* The subject is a male or non-pregnant female between 40 and 75 years of age.
* Patients with a BMI < 35.
* Patients requiring uncemented primary THA, suitable for the use of the uncemented Trident® Hemi HA or Trident® II Clusterhole HA acetabular component in combination with any compatible Stryker femoral stem.
* Patients with no clinical relevant disorders undergoing total hip arthroplasty.
* Patients with a diagnosis of osteoarthritis (OA), avascular necrosis (AVN) or post-traumatic arthritis (TA).
* Patients who are physically and mentally willing and able to comply with postoperative functional evaluation and able to participate in an appropriate rehabilitation schedule.

Exclusion Criteria:

* Patients who are unwilling to cooperate with the study protocol and follow-up schedule.
* Patients who, as judged by the surgeon, are mentally incompetent or are likely to be non-compliant with the prescribed post-operative routine and follow-up evaluation schedule.
* Patients with rheumatoid arthritis hip as well as history of acetabular or femoral osteotomy.
* Patients who had a THA on the contra-lateral side within last 6 months.
* Patients who had or will need lower joint replacement for another joint within 6 month
* Female patients that are pregnant or planning a pregnancy during the course of the study
* Patients who require revision of a previously implanted THA.
* Obese patients where obesity is severe enough to affect subject's ability to perform activities of daily living (body mass index, kg/m2 > 35)
* Patients with active or suspected infection
* Patients with active malignancy
* Patients with a diagnosed systemic disease that would affect the subject's welfare or overall outcome of the study (severe osteoporosis, Paget's disease, renal osteodystrophy) or is immunologically suppressed, or receiving steroids in excess of physiologic dose.
* Patients with a neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device or the patient has a neurological deficit which

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2031-05-11 (Estimated)

PRIMARY OUTCOMES:
Migration, measured by means of RSA | 2 years
  Migration (MTPM in mm) of the prosthesis with respect to the host bone

SECONDARY OUTCOMES:
Migration, measured by means of RSA | 10 years
  Migration (MTPM in mm) of the prosthesis with respect to the host bone
Investigation of clinical performance and patient outcome with EuroQuol-5 dimension (EQ-5D) patient questionnaire | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  The EQ-5D-3L consists of questions covering five dimensions measuring the patient's mobility, self-care, usual activities, pain/discomfort and anxiety/depression, each question with three levels of possible answers and a single index value for health status. Health status has a range from 1 to 100.
Investigation of clinical performance and patient outcome with the Forgotten Joint Score (FJS) patient questionnaire. | 3 months, 1, 2, 5, 7 and 10 years
  The FJS consists of 12 questions and focuses on the patients' awareness of their joint replacement during a range of day to day and recreational activities. The FJS uses a 5-grade Likert scale ranging from "Never" to "Mostly". The score has a range of 0-100.
Investigation of the patients' opinion about their hip and associated problems with HOOS (Hip disability and Osteoarthritis Outcome Score). | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  HOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and hip related Quality of life (QOL). The HOOS uses a 5-grade Likert scale and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Investigation of patient outcome with radiographic analysis | pre-operative, 3 months, 1, 2, 5, 7 and 10 years
  Plain radiographs will be obtained for assessment of fixation of the device.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics Hässleholm-Kristianstad-Ystad, Hässleholm Hospital, Hässleholm, Sweden